CLINICAL TRIAL: NCT07291726
Title: Composite Dietary Antioxidant Index and Metabolic Health in Overweight/Obesity in U.S. Adults: Evidence From NHANES: 2003-2020
Brief Title: Composite Dietary Antioxidant Index and Metabolic Health in Overweight/Obesity in U.S. Adults
Status: Completed | Type: Observational
Sponsor: University-Town Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jiang Peng, Attending Physician, University-Town Hospital of Chongqing Medical University
Other Study IDs: NHANES_CrossSec_2025_01
Record Dates: First submitted 2025-09-29; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Overweight/Obesity; Metabolic Health
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CDAI Q1 (Lowest Quartile)
  Interventions: Other: None (Observational)
- CDAI Q2 (Second Quartile)
  Interventions: Other: None (Observational)
- CDAI Q3 (Third Quartile)
  Interventions: Other: None (Observational)
- CDAI Q4 (Highest Quartile)
  Interventions: Other: None (Observational)

INTERVENTIONS:
Other: None (Observational) — This is an observational study with no active intervention implemented. Its primary aim is to analyze the relationship between the Composite Dietary Antioxidant Index (CDAI) and overweight/obesity, as well as the associated metabolic abnormalities, using the dataset-with no experimental manipulation involved.

SUMMARY:
This cross-sectional study draws on data from the National Health and Nutrition Examination Survey (NHANES) database. The primary objective is to investigate the associations between the Composite Dietary Antioxidant Index (CDAI) and overweight/obesity, as well as the related metabolic abnormalities, among the U.S. general population. By analyzing this large-scale, nationally representative dataset, the investigators seek to generate evidence that can inform public health policies and clinical practice-ultimately contributing to a deeper understanding of population-level health challenges and the development of targeted strategies to address them.

ELIGIBILITY:
Inclusion Criteria:

* Participants with complete data on composite dietary antioxidant index from the NHANES database
* Participants with complete body mass index (BMI) data from the NHANES database
* Individuals aged 18 years and older

Exclusion Criteria:

* Participants with missing key data (composite dietary antioxidant index or BMI)
* Individuals who are pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals from the National Health and Nutrition Examination Survey (NHANES) database. It includes participants aged 18 and above with complete data on dietary antioxidant index and body mass index, representing a nationally representative sample of the U.S. population.
Sampling Method: Probability Sample
Enrollment: 38646 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Overweight/Obesity Assessed by Body Mass Index (BMI) | Baseline: Data collection for calculating BMI occurs during the specific NHANES survey cycle relevant to this study (single - time - point cross - sectional assessment).
  Body Mass Index (BMI) will be calculated as weight (in kilograms) divided by the square of height (in meters). According to the World Health Organization's classification, a BMI of 25.0 - 29.9 kg/m² is considered overweight, and a BMI of 30.0 kg/m² or higher is considered obese. Data on weight and height will be obtained from the NHANES dataset.
Metabolic Phenotype Classification (Metabolically Healthy vs. Unhealthy) Assessed by NCEP ATP III Metabolic Syndrome Components | Baseline: Data on metabolic components for phenotype classification will be collected during the corresponding NHANES survey cycle for this study, reflecting a single-time-point cross-sectional assessment.
  Metabolic phenotypes are classified as metabolically healthy or unhealthy based on the components of metabolic syndrome defined in the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Waist circumference data is not used in this classification due to its high correlation with BMI.
  A participant is defined as metabolically healthy if they have none or only one of the following four metabolic abnormalities: (1) Serum triglycerides (TG) ≥ 150 mg/dL; (2) Serum high-density lipoprotein cholesterol (HDL-C) < 40 mg/dL in men or < 50 mg/dL in women; (3) Fasting glucose ≥ 100 mg/dL or use of hypoglycemic drugs; (4) Blood pressure ≥ 130/85 mmHg or use of antihypertensive drugs.
  A participant is defined as metabolically unhealthy if they have two or more of the above metabolic abnormalities. Relevant data will be retrieved from the NHANES database.

CONTACTS AND LOCATIONS:
Locations (1):
- University Town Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China